CLINICAL TRIAL: NCT04447118
Title: A Phase 3, Randomized, Open-label, Multicenter Study of the Efficacy and Safety of Pyrotinib Versus Docetaxel in Patients With Advanced Non-squamous Non-small Cell Lung Cancer (NSCLC) Harboring a HER2 Exon 20 Mutation Who Progressed on or After Treatment With Platinum Based Chemotherapy
Brief Title: Phase 3 Study of Pyrotinib Versus Docetaxel in Patients With Advanced Non-squamous NSCLC Harboring a HER2 Exon 20 Mutation Who Failed Platinum Based Chemotherapy
Acronym: PYRAMID-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR-BLTN-III-NSCLC
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Non-squamous NSCLC; HER2 Exon 20 Mutation
Keywords: pyrotinib; docetaxel; HER2 Exon 20 Mutation; NSCLC
MeSH Terms: interventions — pyrotinib; Docetaxel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In this study, the Blinded Independent Review Committee (BIRC) will perform a blinded evaluation on the primary endpoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study treatment Arm (Experimental): Pyrotinib maleate tablet, 400 mg, once daily (QD)
  Interventions: Drug: Pyrotinib
- Control Arm (Active Comparator): Docetaxel injection, 75 mg/m2, once every 3 weeks (Q3W)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Pyrotinib — 400 mg, once daily (QD), will be administered with water within 30 minutes after completion of a meal, at approximately the same time each day on a continuous daily dosing schedule, with 21 days as a cycle.
  Other Names: Irene
  Arms: Study treatment Arm
Drug: Docetaxel — 75 mg/m2, once every 3 weeks (Q3W), will be administered by intravenous infusion over 1 hour, with 21 days as a cycle.
  Other Names: Docetaxel injection
  Arms: Control Arm

SUMMARY:
This is a randomized, positive-controlled, open-label, international multicenter, Phase 3 clinical study to compare the efficacy and safety of pyrotinib versus docetaxel in patients with advanced non-squamous NSCLC harboring a HER2 exon 20 mutation who failed platinum based chemotherapy.

DETAILED DESCRIPTION:
150 eligible subjects will be randomized in a 2:1 ratio (Study treatment Arm: Control Arm = 100 : 50 subjects) to receive pyrotinib or docetaxel monotherapy.

Each treatment cycle is defined as 21 days for subjects in both arms. Treatment regimen of pyrotinib (Study treatment Arm): 400 mg/d (QD) oral pyrotinib will be administered within 30 minutes after completion of a meal.

Treatment regimen of docetaxel (Control Arm): 75 mg/m2 (Q3W) of docetaxel will be administered via intravenous infusion.

In this study, crossover treatment is allowed for subjects in Control Arm. Within the specified time window of each cycle, subjects should complete physical examinations, laboratory tests, quality of life questionnaires and other tests to assess the safety and quality of life of the subjects.

During study treatment, tumor radiological assessments will be performed every 6 weeks (42 ± 7 days) in the first 52 weeks and every 12 weeks (84 ± 7 days) thereafter.

After the end of treatment and safety follow-up, all subjects will be followed for survival (every 56 ± 7 days) until death, withdrawal of informed consent, lost to follow-up, or termination of the study (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent which is approved by IRB/EC, willing and able to comply with scheduled treatment, all examinations at study visits, and other study procedures.
* ECOG PS 0-1.
* Have histologically or cytologically confirmed locally advanced or metastatic non-squamous NSCLC disease.
* Before enrollment, a documented confirmed presence of activating mutations in exon 20 of the HER2 gene must be provided. Sufficient tumor tissue samples should be provided to retrospectively confirm the mutation status of the HER2 gene.
* Must have measureable disease per RECIST v1.1.
* For advanced NSCLC, patients must have had progressive disease on or after a platinum based chemotherapy, with or without immune checkpoint inhibitors (PD-1/PD-L1 inhibitors) and/or anti-angiogenic drugs. No more than 2 prior lines of systemic therapy are allowed.
* The laboratory test values must meet the following standards to manifest that the functional level of important organs/systems meets the requirements.
* Female patient of childbearing potential (WOCBP) and male patient whose - partner is WOCBP must agree to use effective contraception method during the study period.

Exclusion Criteria:

* Malignant tumors with other pathological types.
* Medical history of other active malignancies within last 5 years.
* Subjects with active CNS metastases.
* Previously treated with targeted drugs for HER2 gene mutations,or previously treated with docetaxel.
* Prior to the first dose of study treatment, patients with severe effusions with clinical symptoms, severe cardiac disease, or severe infection.
* Prior to the first dose of study treatment, patients with diseases or special conditions that affect drug administration and absorption.
* Congenital or acquired immunodeficiency.
* History of allergy to the study drugs or components.
* Prior to the first dose of study treatment, or during the study period, patients receive or are anticipated to receive continuous strong CYP3A4 inducers or inhibitors, P-gp inhibitors, or medications that are known to cause QT/QTc prolongation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 26 months
  Time from the date of randomization to the date of first disease progression documented by BIRC according to the RECIST v1.1 or death for any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall survival (OS) | 36 months
  Time from the date of randomization to death for any cause.
Objective response rate (ORR) | 26 months
  Assessed by BIRC and investigator according to the RECIST v1.1.
Disease control rate (DCR) | 26 months
  Assessed by BIRC and investigator according to the RECIST v1.1.
Duration of response (DoR) | 26 months
  Assessed by BIRC and investigator according to the RECIST v1.1.
Time to tumor progression (TTP) | 26 months
  Assessed by BIRC and investigator according to the RECIST v1.1.
Progression-free survival 2(PFS2) | 36 months
  Assessed by investigator according to the RECIST v1.1, or death for any cause, whichever comes first.
Patient reported outcome (PRO) using EORTC QLQ-C30 | 26 months
  Symptoms related to NSCLC,
Patient reported outcomes (PRO) using the QLQ-LC13 | 26 months
  Symptoms related to NSCLC
Plasma concentrations of pyrotinib | 26 months
  Pharmacokinetics (PK) of pyrotinib
AEs and SAEs | 26 months
  Judged in accordance with NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi, MD,PhD, Study Director — Jiangsu Hengrui Pharmaceutical Co., Ltd.
Locations (102):
- United States (11):
  - University of California - Irvine Medical Center, Orange, California
  - University of California (UC) Davis Comprehensive Cancer Center, Sacramento, California
  - Innovative Clinical Research Institute, Whittier, California
  - Florida Cancer Specialists South Divisio, Fort Myers, Florida
  - Florida Cancer Specialists North Divisio, St. Petersburg, Florida
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Summit Cancer Centers - North Spokane, Spokane, Washington
- Australia (5):
  - Royal North Shore Hospital, St Leonards, Saint Leonards
  - Border Medical Oncology, Albury
  - St Vincent's Hospital Melbourne, Fitzroy
  - Sir Charles Gairdner Hospital, Nedlands
  - Calvary North Adelaide Hospital, North Adelaide
- Belgium (3):
  - Antwerp University Hospital (UZA), Edegem
  - University Hospital Gent, Ghent
  - University Hospital (UZ) Leuven, Leuven
- China (31):
  - the Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - beijing chest hospital,Capital medical university, Beijing, Beijing Municipality
  - Peking university Cancer Hospital, Beijing, Beijing Municipality
  - The second affiliated hospital of ChongQing medical university, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Cangzhou Hospital of Integrated Tcm-Wm.Hebei, Cangzhou, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - First Affiliated Hospital of ZhengzhouUniversity, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei cancer hospital WardII, Wuhan, Hubei
  - Hunan Cancer Hospital & The Affiliated Cancer Hospital of Xiangya School of Medicine, Central South University, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Subei People's Hospital of Jiangsu Province, Yangzhou, Jiangsu
  - The Second Affiliated of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The affiliated hospital of inner mongolia medical univerity, Hohhot, Neimenggu
  - Shandong Cancer Hospital Affiliated to Shandong University, Jinan, Shandong
  - Shanghai Pulmonary Hospital, Tongji University, Shanghai, Shanghai Municipality
  - Fudan University Cancer hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - SiChuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - The Second People's Hosipital of Yibin, Yibin, Sichuan
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Yunnan Provincial Cancer Hospital, Kunming, Yunnan
  - Sir Run Run Shaw Hospital ZheJiang University School Of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital，ZheJiang University, Hangzhou, Zhejiang
  - ZheJiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
- France (6):
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier Intercommunal Creteil, Créteil
  - AP-HM - Hôpital Nord, Marseille
  - Hopital Bichat - Claude Bernard - AP-HP, Paris
  - CHRU Strasbourg, Strasbourg
  - CHU Toulouse - Hopital Larrey, Toulouse
- Germany (5):
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Uniklinikum Giessen und Marburg, Giessen
  - Klinikverbund Kempten-Oberallgäu gGmbH, Kempten
  - POIS Leipzig GbR, Leipzig
  - Pius-Hospital Oldenburg, Centre of Radiotherapy and Medical Oncology, Dept. Medical Oncology, Oldenburg
- Italy (5):
  - Centro Riferimento Oncologico - Aviano, Aviano
  - Azienda Ospedaliero Universitaria Policlinico G. Rodolico-San Marco - Presidio Ospedaliero G. Rodolico, Catania
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori, Meldola (FC)
  - Istituto Europeo di Oncologia, Milan
  - ASST dei Sette Laghi-Ospedale di Circolo e Fondazione Macchi di Varese, Varese
- Poland (4):
  - Centrum Onkologii KOMED, Konin
  - Salve-Medica, Lodz
  - Instytut Genetyki i Immunologii GENIM, Lublin
  - Med Polonia Sp. z o.o., Poznan
- Russia (6):
  - Petrov National Medical Research Center of Oncology, Saint Petersburg, Sankt-Peterburg
  - Arkhangelsk Clinical Oncological Dispensary, Arkhangelsk
  - JSC Group of companies Medsi, Moscow
  - Clinical hospital RZD-Medicine of St. Petersburg, Saint Petersburg
  - Eurocityclinic LLC, Saint Petersburg
  - Saint-Petersburg Clinical Research Center of Specialized Types of Medical Care (Oncology), Saint Petersburg
- South Korea (7):
  - Seoul National University Bundang Hospital, Seoul, Bundang
  - Ajou University Hospital, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (9):
  - Hospital Germans Trias i Pujol, Barcelona, Badalona
  - Hospital Universitario Vall d'Hebron, Barcelona, Badalona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario Virgen del Rocio, Seville
  - Instituto Valenciano de Oncologia, Valencia
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital (CGMHLK), Taoyuan
- Turkey (Türkiye) (7):
  - Baskent University Adana Application and Research Center, Adana
  - Ankara Sehir Hastanesi, Ankara
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Izmir Medical Park Hospital, Izmir
  - Gulhane Training and Research Hospital, Keçiören
  - Necmettin Erbakan University Selcuklu Faculty of Medicine, Konya
  - Trakya University Medical Faculty, Merkez

IPD SHARING:
Plan to Share IPD: No